CLINICAL TRIAL: NCT05157763
Title: An Open-Label Study to Evaluate the Safety and Efficacy of EscharEx (EX-02) in the Treatment of Basal Cell Carcinoma
Brief Title: A Study to Evaluate the Safety and Efficacy of EscharEx (EX-02) in the Treatment of Basal Cell Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MediWound Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MW2020-11-26
Record Dates: First submitted 2021-05-06; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Superficial Basal Cell Carcinoma; Nodular Basal Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EscharEx 5% (Experimental): The powder of EX-02 (4 g per vial) should be reconstituted with 10 ml water for injection (WFI) to obtain 5% EX-02 gel. The EX-02 powder and the WFI are to be mixed up to 15 min prior to use. EX-02 5% gel will be topically applied in a thick layer of 2-3 mm on the lesion surface including margin of 5-10 mm for 8-12 hours (preferable over-night) and covered with an occlusive dressing. A new vial should be used for each application. Each patient will be treated with 7 applications.
  Interventions: Drug: EscharEx 5% (EX-02 formulation)

INTERVENTIONS:
Drug: EscharEx 5% (EX-02 formulation) — EX-02 5% will be topically applied in a thick layer of 2-3 mm on the lesion surface for 8-12 hours including 5-10 mm margins and covered with an occlusive dressing. A new vial should be used for each application. Each patient will be treated with 7 applications.
  Other Names: EX-02 5%

SUMMARY:
This study will be a multicenter, prospective, open label, one-arm study intended to assess the Safety and Efficacy of EscharEx (EX-02) in the treatment of Basal Cell Carcinoma.

In patients with one primary superficial or nodular basal cell carcinoma lesion with a diameter of 5-10mm (Histologically confirmed BCC) located on the trunk or upper extremities (not including the hands), with well-defined borders and no previous radiation therapy.

DETAILED DESCRIPTION:
32 patients are planned to be enrolled into the study from 2-4 US sites. This study will be an Open-Label Study where all patients will be treated with the investigational product EX-02.

Enrollment will be conducted in 2 stages. In the first stage, a group of sixteen (16) patients will be enrolled and treated as detailed below for group 1. Safety results from the first group of patients will be evaluated by the sponsor and by the DSMB. Based on the safety results and DSMB recommendations, the second group of patients will include additional 16 patients that will be enrolled and treated, as detailed below for group 2. All patients will undergo complete surgical excision at the end of the 8 weeks post treatment period and will be followed up until complete clearance is confirmed by biopsy and the wound is closed.

Each patient will go through the following periods during the trial:

1. Screening and enrollment period (up to 2 weeks, visit#1):

   Screening and enrollment duration will be up to 2 weeks and will include the following:

   signing informed consent, recording demographics, medical history and concomitant medications, vital signs, physical examination, lesion photography and assessments, and shave biopsy. Only patients with histologically confirmed BCC can be enrolled and start treatment.
2. Treatment Period (1-3 weeks, 10-14 visits- visits#2-15)

   Group 1: 16 patients- 8 patients with superficial BCC and 8 patients with nodular BCC will undergo 7 treatment applications, once every other day (2 weeks).

   Group 2: Based on safety results of stage 1 and following DSMB review and recommendations, 16 additional patients (8 patient with superficial BCC and 8 patients with nodular BCC) will undergo 7 daily applications. In case of tolerability issues a rescue therapy of either 7 applications every other day (same as in group 1) or 1 day of drug holiday after which daily treatment will continue, will be allowed as needed.

   In both groups, EX-02 5% will be topically applied on the lesion's surface including a margin of 5-10mm, for 8-12 hours each application. All pre application assessments and applications s will be performed at the clinic. Dressing removal will be completed by the patient (by a family member/caregiver) at the patient's home. Between applications, the lesion will be covered by hydrocolloid dressing (applied by the patient or by a family member/caregiver). The treatment area including the skin around the lesion will be photographed before each application at the clinic and assessment of AEs will be performed by the investigator before application and post dressing removal.

   This period will include 10 on-site visits, 7 visits for pre application assessments and drug application (visits# 2, 4, 6, 8,10, 12, 14) and 3 on-site visits for post dressing removal and assessments. The following three (3) post dressing removal visits will be performed at the clinic: after first application (post dressing removal) (visit#3), after second application (post dressing removal) (visit#5) and after last application (post dressing removal) (Visit#15). Additional 4 visits post dressing removal (visits#7, 9, 11 and 13) are optional and will be completed only if needed per PI discretion. These optional visits, if performed, can be performed either at the clinic or remotely (by an IRB approved HIPAA compliance telecommunication). Local lab tests will be obtained on visits#1(screening) and visit#15.
3. Post Treatment period (8 weeks, 4 bi-weekly remote or on site visits, visit#16-19):

   Post completion of treatment course, the raw bed and the surrounding skin will be treated toward healing of the skin by Vaseline petrolatum or Aquaphor. Once in 2 weeks the treated area will be photographed, the healing status of the wound and adverse events will be assessed. Assessments on first 3 bi-weekly visits, visit#16- 18 will be performed either on site or remotely (via IRB approved, HIPAA compliance telecommunication), based on physician discretion. The 4th bi-weekly visit i.e. Visit #19 will be performed on site. At the end of the 8 weeks post treatment period, on the 4th bi-weekly visit (visit#19), all patients will undergo complete excision, including a lesion margin of 4-5 mm. The specimen will be sent to dermapathologist for histological clearance examination.
4. Follow Up (until complete clearance and wound closure is achieved, at least one visit):

During the follow up stage, patients will be followed and treated with standard of care. Follow up visit # 20 will be performed once biopsy results are available (from the excision performed on visit#19). Results will be recorded in the eCRF. In cases that margins are not clear, patients will undergo additional excisional procedure per standard of care. Histological results from any additional procedure will be recorded. In cases that margin are clear but additional procedure for wound closure is required, the procedure will be recorded. AEs will be monitored until complete clearance of margins is histologically confirmed and until wound is assessed as closed (and sutured were removed).

The total duration of the study for each participating subject is approximately 14-17 weeks: Screening periods (1-2 weeks) + Treatment (1-3 weeks) + Follow up post treatment and histopathology 8 weeks post treatment + Follow up post-surgical excision (approximately 4 weeks- until wound closure).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria- Patient level

1. Male or female greater than age 18,
2. Patients with one primary superficial or nodular basal cell carcinoma lesion (Histologically confirmed BCC) located on the trunk or upper extremities (not including the hands), with well-defined borders and no previous radiation therapy.
3. Lesion is present for no longer than 4 years.
4. Lesion with a diameter of 5-10mm,
5. Patient and/or legally authorized representative (LAR) understands the nature of the procedure, is able and willing to adhere to the protocol regimen, and able to provide a written informed consent prior to any study procedure.

Exclusion Criteria:

Exclusion Criteria- Patient level

1. Evidence of Gorlin syndrome, neoplastic diseases (except actinic lesions), metastatic tumor or tumor with high probability of metastatic spread,
2. Other malignant cancers (non BCC) of the skin at the lesion's site,
3. Morphea-type basal cell carcinoma (MBCC) at the lesion's site (per biopsy report),
4. Any signs of infection at the lesion site including purulent discharge, tissue abscess, erysipelas, cellulitis, etc.,
5. Patients with any dermatological disease in the target lesion site or surrounding area (not including chronic actinic damage in the surrounding area),
6. History of allergy or atopic disease or a known sensitivity to pineapples, papaya, bromelain or papain, as well as known sensitivity to latex proteins (known as latex-fruit syndrome), bee venom or olive tree pollen,
7. Patients undergoing renal or peritoneal dialysis,
8. Any condition that would preclude safe participation in the study, e.g. evidence of significant or unstable cardiovascular, pulmonary, liver, hematological, immunological, or any immediate life threatening condition,
9. Concurrent acute injury or disease that might compromise the patient's welfare or the participation in the study,
10. Current (within last 12 months) severe alcohol or drug use disorder
11. Pregnant women (positive blood or urine pregnancy test) or nursing mothers,
12. Exposure to investigational intervention within 4 weeks prior to enrolment, or anticipated participation in another investigational drug trial or other intervention trial, while enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent AEs (TEAEs) and serious TEAEs (STEAEs). | Through study completion - an average of 16 weeks
  All adverse events (AEs) will be listed. Adverse events records will include notification whether the AE is local and occurs near or in the target lesion. The AEs will be listed as counts and percentages by System Organ Class (SOC), Preferred Term (PT), severity, and time of onset. Serious Adverse Events will be analyzed in the same way as AEs
Vital signs - proportion of patients with abnormal clinical significant measurements | Up to completion of treatment period - up to 5 weeks
  Assessed pre 2nd, pre 5th application and post last application
Pain assessments- Proportion of patients with clinical significant elevation in NPRS score | Up to completion of treatment period - up to 5 weeks
  Assesed pre 2nd, pre 5th application and post last application compared with pre 1st application
Proportion of subjects discontinuing a treatment due to TEAEs, assessed over the entire course of the treatment. | Up to completion of treatment period - up to 5 weeks
  This proportion will be calculated, together with its 95% confidence interval based on the binomial distribution.
Proportion of subjects that requested to discontinue the treatment | Up to completion of treatment period - up to 5 weeks
  This will be assessed over the entire course of the treatment and will be calculated, together with its 95% confidence interval based on the binomial distribution

SECONDARY OUTCOMES:
Proportion of patients who reached complete histological clearance at the end of the post treatment period. | Up to 13 weeks
  biopsy will be taken 8 weeks post completion of treatment. The proportion of patients who reached complete histological clearance at the end of the post treatment period, together with its 95% confidence interval based on the binomial distribution.
Proportion of patients who reached complete clearance at the end of the post treatment period, as clinically assessed prior to surgical removal. | Up to 13 weeks
  The proportion of patients who reached complete histological clearance as assessed by the investigator at the end of the post treatment period, prior to the excisional biopsy, together with its 95% confidence interval based on the binomial distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Lior Rosenberg, Prof., Study Director — MediWound Ltd
Locations (3):
- United States (3):
  - Center for Clinical and Cosmetic Research, Aventura, Florida
  - Moore Clinical Research, Inc., Brandon, Florida
  - Center for Clinical Studies, LTD. LLP, Webster, Texas

IPD SHARING:
Plan to Share IPD: No